CLINICAL TRIAL: NCT06492850
Title: A Phase I/II Dose-escalation and Dose-expansion Study to Evaluate the Safety and Efficacy of FT-002 Subretinal Injection in Subjects With RPGR Gene Mutation-associated X-linked Retinitis Pigmentosa.
Brief Title: Gene Therapy for RPGR Gene Mutation-associated X-linked Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT002-C101
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: X-Linked Retinitis Pigmentosa (XLRP)
Keywords: X-Linked Retinitis Pigmentosa (XLRP); FT-002

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FT-002 dose 1 (Experimental): Low dose FT-002
  Interventions: Genetic: FT-002
- High dose FT-002 (Experimental): High dose FT-002
  Interventions: Genetic: FT-002

INTERVENTIONS:
Genetic: FT-002 — Intraocular injection of a single dose

SUMMARY:
The aim of this study was to evaluate the safety, tolerability, and efficacy of one-time subretinal injection of FT-002 in male subjects (8-45 years of age) with RPGR (Retinitis Pigmentosa GTPase Regulator) gene mutation-associated X-linked retinitis pigmentosa, of XLRP. This study includes Phase I (dose escalation phase) and Phase II (dose expansion phase).

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are willing and able to follow study procedures including scheduled visits, treatment plan, and laboratory tests, and sign a written informed consent form;
* Age: Phase I dose escalation stage, 18-45 years old male (including boundary value) at the time of signing the ICF; Phase II dose extension stage, males 8-45 years old (including boundary values) at the time of signing the ICF;
* Clinically diagnosed XLRP, the main symptoms include but are not limited to night blindness, visual field loss, vision loss, etc.;

Exclusion Criteria:

* Have other retinal degenerative diseases, such as retinal degeneration caused by other known Inherited retinal disease gene variants or previously received an gene therapy product.

Ages: 8 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerance of FT-002 | from FT-002 administration through up to 1 years
  Incidence and severity of AEs

SECONDARY OUTCOMES:
To evaluate the efficacy of FT-002 | from FT-002 administration through up to 1 years
  Changes in visual sensitivity /FST/BCVAfrom baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ruifang Sui, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No